CLINICAL TRIAL: NCT02769858
Title: The Effects of Light Therapy on Circadian Rhythms, Sleep, and Mood in Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Leslie Swanson, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G016030
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Light Therapy (Experimental): Participants will use commercially-available light therapy glasses (Re-Timer) daily for 60 minutes for five weeks.
  Interventions: Device: Light therapy

INTERVENTIONS:
Device: Light therapy — Light therapy glasses
  Other Names: Re-Timer

SUMMARY:
The proposed study aims to establish the feasibility of light therapy for postpartum depression delivered via Re-Timer, demonstrate its preliminary efficacy, and illuminate relationships between circadian shifts and mood changes using a novel, home-based circadian biomarker assessment paradigm (salivary dim light melatonin onset; DLMO).

ELIGIBILITY:
Inclusion Criteria:

* Within 6 months postpartum
* Meet DSM-V diagnostic criteria for MDD
* Score ≥ 20 on the Structured Interview Guide for the Hamilton Depression Rating Scale-Seasonal Affective Disorder version (SIGH-SAD).

Exclusion Criteria:

* current diagnosis of bipolar disorder, posttraumatic stress disorder, schizophrenia or psychosis, dissociative disorders, eating disorder, obsessive-compulsive disorder, somatic symptom and related disorders, substance use disorder, panic disorder, agoraphobia per DSM-V
* past history of mania/hypomania,
* chronic medical conditions associated with depression (e.g., thyroid conditions)
* ocular or retinal pathology
* history of seizures or epilepsy
* color blindness
* Lupus
* currently taking an antibiotic, medication that contains hydrochlorothiazide, or isotretinoin (Accutane).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Swanson, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swanson LM, Burgess HJ, Zollars J, Todd Arnedt J. An open-label pilot study of a home wearable light therapy device for postpartum depression. Arch Womens Ment Health. 2018 Oct;21(5):583-586. doi: 10.1007/s00737-018-0836-z. Epub 2018 Mar 30. PMID 29603017

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Light Therapy
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Light Therapy
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Score of the Hamilton Depression Rating Scale-Seasonal Affective Version (SIGH-SAD) at 5 Weeks
Description: Clinician-rated depression symptom severity measure; Hamilton Depression Rating Scale-Seasonal Affective Version (SIGH-SAD) (29 item version) measures depressive symptoms on a continuous scale. Higher scores indicate worse outcomes. Scores can range from 0 -73, where 0 means no depression, and 73 is the greatest possible depression. Generally scores of 20 or higher represent clinical depression
Time Frame: After five weeks of light therapy
Measure: Mean (Standard Deviation); unit: SIGH-SAD score
Arm/Group | Light Therapy
Number analyzed (Participants) | 8
SIGH-SAD score
  Pre-treatment | 24.75 (4.83)
  Post-treatment | 12.88 (7.88)
Statistical Analysis 1: Comparison: Light Therapy; Test type: Other; p = .001, t-test, 2 sided

2. Primary Outcome: Change From Baseline Score of the Edinburgh Postnatal Depression Scale (EPDS) at 5 Weeks
Description: Self-report of depression symptoms. The Edinburgh Postnatal Depression scale is scored from 0 to 30 where 0 is no depression and 30 is most severe depression.
Time Frame: After five weeks of light therapy
Measure: Mean (Standard Deviation); unit: EPDS score
Arm/Group | Light Therapy
Number analyzed (Participants) | 8
EPDS score
  Pre-Treatment (EPDS | 12.75 (4.2)
  Post-Treatment (EPDS) | 7.75 (7.50)
Statistical Analysis 1: Comparison: Light Therapy; Test type: Other; p = .019, t-test, 2 sided

3. Primary Outcome: Change From Baseline Time of Dim Light Melatonin Onset (DLMO) at 5 Weeks
Description: Onset of melatonin in dim light conditions as measured in saliva (also called DLMO) Time of DLMO is measured in clock time, so a positive number in change would represent a later onset of melatonin and a negative number represents an earlier onset of melatonin
Time Frame: After five weeks of light therapy
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Light Therapy
Number analyzed (Participants) | 8
minutes | -6 (20)
Statistical Analysis 1: Comparison: Light Therapy; Test type: Other; p = .502, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Light Therapy
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Light Therapy (N=10)
Headache (Nervous system disorders) | 5
Irritability (Psychiatric disorders) | 4
Eyestrain (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No